CLINICAL TRIAL: NCT00006122
Title: Gemtuzumab Ozogamicin (CMA-676) Followed or Not by Intensive Chemotherapy as Initial Treatment for Elderly Patients With Acute Myeloid Leukemia: An EORTC-LG Pilot Phase II Study
Brief Title: Gemtuzumab Ozogamicin With or Without Chemotherapy in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-06993; EORTC-06993-AML-15
Record Dates: First submitted 2000-08-03; First posted 2004-02-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Cytarabine; Etoposide; Gemtuzumab; Idarubicin; Mitoxantrone

INTERVENTIONS:
Drug: cytarabine
Drug: etoposide
Drug: gemtuzumab ozogamicin
Drug: idarubicin
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy uses different ways to stop cancer cells from dividing so they stop growing or die. Combining gemtuzumab ozogamicin with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of gemtuzumab ozogamicin with or without chemotherapy in treating older patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility, toxicity, and antileukemic activity of gemtuzumab ozogamicin (CMA-676) with or without mitoxantrone, etoposide, cytarabine, and idarubicin in elderly patients with acute myeloid leukemia.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (standard risk, defined as age 61-75 and WHO performance status 0-1 vs poor risk, defined as over 75 years and WHO performance status 0-2 OR under 76 years and WHO performance status 2). Frontline therapy: Patients receive gemtuzumab ozogamicin IV over 2 hours on days 1 and 15. Stratum I (Standard risk patients): Patients with disease progression at any time during frontline therapy may begin induction therapy immediately. Induction therapy begins 7-10 days after response assessment regardless of response and in the absence of unacceptable toxicity. Stratum II (Poor risk patients): Patients experiencing complete remission with or without platelet recovery will begin consolidation therapy within 4-8 weeks of response assessment in the absence of unacceptable toxicity. Stratum I Induction therapy: Patients receive mitoxantrone IV over 30 minutes on days 1, 3 and 5; etoposide IV over 1 hour on days 1-3; and cytarabine IV continuously on days 1-7. Patients experiencing partial response are given a second induction therapy course. Patients experiencing complete remission with or without platelet recovery after 1 or 2 induction courses begin consolidation therapy within 4-8 weeks of response assessment in the absence of unacceptable toxicity. Consolidation therapy: Patients receive idarubicin IV on days 1, 3 and 5; etoposide IV over 1 hour on days 1-3; and cytarabine IV continuously on days 1-5. Stratum II Consolidation therapy: Patients receive gemtuzumab ozogamicin IV over 2 hours on day 1 and then 1-3 months later. Patients are followed monthly for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 45-82 (28-49 for stratum I, and 17-33 for stratum II) patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of primary or secondary acute myeloid leukemia (AML) Previously untreated At least 20% marrow blasts AML after myelodysplastic syndrome allowed No leukemia after other myeloproliferative diseases No acute promyelocytic leukemia (M3) or blastic phase chronic myelogenous leukemia No active CNS leukemia

PATIENT CHARACTERISTICS: Age: 61 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics White blood count no greater than 30,000/mm3 unless reducible to less than 30,000/mm3 by a maximum of 7 days of hydroxyurea Hepatic: Bilirubin no greater than 3 times upper limit of normal (ULN) Renal: Creatinine no greater than 3 times ULN Cardiovascular: No severe heart failure that would preclude study Pulmonary: No severe lung failure that would preclude study Other: No other concurrent malignancies No active uncontrolled infection No concurrent severe neurological or psychiatric disease No psychological, familial, sociological or geographical condition that would preclude compliance with study HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior humanized monoclonal antibody therapy Chemotherapy: Up to 7 days of prior hydroxyurea allowed At least 24 hours since prior hydroxyurea No other prior chemotherapy for AML Endocrine therapy: No more than 7 days of prior corticosteroids No other prior endocrine therapy Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2000-06; Primary Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Amadori, MD, Study Chair — Ospedale Sant' Eugenio
Locations (18):
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Belgium (3):
  - A.Z. St. Jan, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Sart-Tilman, Liège
- University Hospital Rebro, Zagreb, Croatia
- France (3):
  - Hopital Edouard Herriot, Lyon
  - Hotel Dieu de Paris, Paris
  - Hopital Necker, Paris
- Germany (2):
  - Medizinische Klinik und Poliklinik, Heidelberg
  - Eberhard Karls Universitaet, Tübingen
- Italy (5):
  - Ospedale Generale Regionale, Bolzano
  - Ospedali Riuniti, Reggio Calabria
  - Ospedale San Eugenio, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Netherlands (3):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen

REFERENCES:
- [Background] Seedhouse CH, Grundy M, White P, Li Y, Fisher J, Yakunina D, Moorman AV, Hoy T, Russell N, Burnett A, Pallis M; National Cancer Research Network. Sequential influences of leukemia-specific and genetic factors on p-glycoprotein expression in blasts from 817 patients entered into the National Cancer Research Network acute myeloid leukemia 14 and 15 trials. Clin Cancer Res. 2007 Dec 1;13(23):7059-66. doi: 10.1158/1078-0432.CCR-07-1484. PMID 18056183
- [Result] Amadori S, Suciu S, Willemze R, et al.: Up-front window trial of gemtuzumab ozogamicin (GO) in previously untreated elderly patients with AML: an EORTC leukemia group study. [Abstract] Blood 104 (11): A-877, 2004.
- [Result] Amadori S, Suciu S, Willemze R, Mandelli F, Selleslag D, Stauder R, Ho A, Denzlinger C, Leone G, Fabris P, Muus P, Vignetti M, Hagemeijer A, Beeldens F, Anak O, De Witte T; EORTC leukemia group; GIMEMA leukemia group. Sequential administration of gemtuzumab ozogamicin and conventional chemotherapy as first line therapy in elderly patients with acute myeloid leukemia: a phase II study (AML-15) of the EORTC and GIMEMA leukemia groups. Haematologica. 2004 Aug;89(8):950-6. PMID 15339678